CLINICAL TRIAL: NCT00592137
Title: Calcium, Dairy, and Body Fat in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Connie Weaver/Professor and Head of Department, Department of Foods and Nutrition, Purdue University
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DK66108 (completed); 5R01DK066108 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Energy Metabolism
Keywords: calcium carbonate; obesity; dairy; energy expenditure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C (Placebo Comparator): During one three week session of a controlled diet subjects will receive a smoothie based on soy protein two times per day that does not contain any additional calcium
  Interventions: Dietary Supplement: C (smoothies based on soy protein containing no additional calcium)
- B (Active Comparator): During one three week period half of the participants will receive two smoothies per day based on soy protein that contain 650 mg Ca as calcium carbonate
  Interventions: Dietary Supplement: B (smoothies based on soy protein containing calcium)
- A (Active Comparator): During one three week session subjects will receive two smoothies per day based on dairy protein containing 650 mg calcium
  Interventions: Dietary Supplement: A (smoothies based on dairy protein containing calcium)

INTERVENTIONS:
Dietary Supplement: C (smoothies based on soy protein containing no additional calcium) — Two smoothies per day based on soy protein containing no additional calcium
  Arms: C
Dietary Supplement: B (smoothies based on soy protein containing calcium) — Two smoothies daily based on soy protein containing 650 mg calcium as calcium carbonate
  Arms: B
Dietary Supplement: A (smoothies based on dairy protein containing calcium) — Two smoothies daily based on dairy protein containing 650 mg calcium
  Arms: A

SUMMARY:
Lifestyle choices,including diet,are conducive to healthy body weights in children. Dairy products and calcium supplementation have been associated with moderation of body weight and body fat. This study was designed to test the following hypotheses with overweight and obese adolescents consuming a controlled diet:

* Dietary calcium supplementation as calcium carbonate or dairy calcium modulates energy balance in adolescents.
* Increased calcium in the diet of adolescents will increase fecal fat excretion and thereby decrease fat absorption.
* Calcium and dairy product supplementation will increase lipid oxidation resulting in an increase in energy expenditure.

DETAILED DESCRIPTION:
Subjects will consume a controlled diet containing 800 mg calcium for two three week periods. During one period they will also receive a frozen ice cream like product (smoothie) twice a day based on soy protein that contains no additional calcium. During the other period they will receive a similar product twice a day based on either dairy protein that contains 650 mg calcium or based on soy protein that contains 650 mg calcium as calcium carbonate

ELIGIBILITY:
Inclusion Criteria:

* Over weight (>85th percentile BMI for age)

Exclusion Criteria:

* > 180% of ideal body weight for height
* Malabsorptive disorders
* Bone disease
* Liver disease
* Kidney disease
* Anemia
* Smoking or illegal drugs
* Oral contraceptives
* Pregnancy
* Medications that influence calcium metabolism

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2004-04; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Energy balance will be calculated by quantitating the kilocalories represented by the following components: dietary intake, excreta, physical activity, resting energy expenditure, thermic effect of food, and thermogenesis. | After equilibration on a controlled diet for one week, measurements will be taken over an additional two week period.

SECONDARY OUTCOMES:
Serum biochemical measures of calcium metabolism (PTH, Vitamin D, and calcium) | Serial meausures over a 10 hour period following a meal containing calcium from the placebo, dairy or calcium carbonate supplement
Calcium retention | Two weeks on a controlled diet following one week of equilibration on the same diet

CONTACTS AND LOCATIONS:
Overall Officials: Connie Weaver, PHD, Principal Investigator — Department Foods and Nutrition, Purdue University; Berdine R Martin, PhD, Study Director — Department Foods and Nutrition, Purdue University
Locations (1):
- Department of Foods and Nutrition, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Weaver CM, Campbell WW, Teegarden D, Craig BA, Martin BR, Singh R, Braun MM, Apolzan JW, Hannon TS, Schoeller DA, DiMeglio LA, Hickey Y, Peacock M. Calcium, dairy products, and energy balance in overweight adolescents: a controlled trial. Am J Clin Nutr. 2011 Nov;94(5):1163-70. doi: 10.3945/ajcn.110.010264. Epub 2011 Sep 14. PMID 21918216
- [Derived] Singh R, Martin BR, Hickey Y, Teegarden D, Campbell WW, Craig BA, Schoeller DA, Kerr DA, Weaver CM. Comparison of self-reported, measured, metabolizable energy intake with total energy expenditure in overweight teens. Am J Clin Nutr. 2009 Jun;89(6):1744-50. doi: 10.3945/ajcn.2008.26752. Epub 2009 Apr 22. PMID 19386746